CLINICAL TRIAL: NCT01127906
Title: A Randomized, Double-Blind, Double-Dummy, Placebo And Active Comparator Controlled 4-Period Cross-Over Study To Assess The Effect Of PF-04531083 On Heat Pain In The UVB-Induced Pain Model In Healthy Volunteers
Brief Title: Study To Assess The Effect Of PF-04531083 On Heat Pain In Healthy Volunteers With Ultraviolet Light Sensitized Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: B1351003
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2010-09-23 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Healthy Volunteers; cross-over; randomized; placebo and active controlled; heat pain; UVB-Induced pain model
MeSH Terms: interventions — Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Randomized cross-over sequence (Other): Randomized unbalanced sequence of incomplete block design with replicates within sequence
  Interventions: Drug: PF-04531083 100mg; Drug: PF-04531083 2000mg; Drug: Placebo suspension; Drug: Placebo tablet; Drug: Oxycodone 20mg

INTERVENTIONS:
Drug: PF-04531083 100mg — Oral PF-04531083 100mg suspension single dose
Drug: PF-04531083 2000mg — Oral PF-04531083 2000mg suspension single dose
Drug: Placebo suspension — Oral Placebo suspension (matched to PF-04531083 suspension)
Drug: Placebo tablet — Oral Placebo tablet (matched to Oxycodone)
Drug: Oxycodone 20mg — Oral Oxycodone 20mg (Oxycontin) controlled release formulation

SUMMARY:
PF-04531083 has been shown to reduce the amount of heat pain experienced by rats with skin that has been sensitized to heat by ultraviolet light. This study is designed to see if this is also true in man.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.
* Body mass index between 17.5 - 30.5 kg/m2 and body weight greater than 50 kg.

Exclusion Criteria:

* Subjects that have any condition possibly affecting drug absorption (eg, gastrectomy).
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* Subjects with inadequate cardiac function (ECG demonstrating prolonged QTc interval at screening).
* Subjects with inadequate or excessive sensitivity to UVB light.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To assess the effect of PF-04531083 by using the Heat Pain Tolerance Threshold in the area of UVB-induced erythema (HPTTu) endpoint at 2, 4, 6 and 24 hours. | 24 hours

SECONDARY OUTCOMES:
Heat Pain Perception Threshold in the area of UVB-induced erythema (HPPTu) at 2, 4, 6 and 24 hours. | 24 hours
Heat Pain Perception Threshold on control skin (HPPTc) at 2, 4, 6 and 24 hours | 24 hours
Summary of plasma concentrations of PF-04531083 | 24 hours
Exploratory colorimetric data collected from baseline and MED test exposure areas | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Brussels, Belgium

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1351003&StudyName=Study%20To%20Assess%20The%20Effect%20Of%20PF-04531083%20On%20Heat%20Pain%20In%20Healthy%20Volunteers%20With%20Ultraviolet%20Light%20Sensitized%20Skin